CLINICAL TRIAL: NCT00174408
Title: Growth Hormone Treatment in Short Children Born Small for Date (Genotonorm)
Brief Title: Treatment Of Children With Short Stature At An Age Of 3-7 Years Who Were Born Small For Gestational Age
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 89-041; A6281048
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2007-05-03 (Estimated); Status verified 2007-05

CONDITIONS: Growth Disorders
MeSH Terms: conditions — Growth Disorders | interventions — Human Growth Hormone

INTERVENTIONS:
Drug: Genotropin

SUMMARY:
The primary objective is to evaluate, if Genotonorm (Genotropin) increases linear growth in short children born SGA. Safety of the drug is a main objective as well. The growth promoting effect of two different dosages is compared. The effect of long-term treatment on final height is evaluated (according to several amendments)

ELIGIBILITY:
Inclusion Criteria:

* Birth length below -2 SD
* Height at start below - 2 Sd

Exclusion Criteria:

* Any endocrine or chronic disease
* Any known syndrome with short stature

Ages: 3 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 110
Dates: Start 1990-03; Study Completion 2005-02

PRIMARY OUTCOMES:
Height, height velocity

SECONDARY OUTCOMES:
Side effects

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer